CLINICAL TRIAL: NCT00612196
Title: A Randomised, Phase I, Single Dose, Placebo-Controlled, Dose Escalation Study of TB-402, A Monocloncal Antibody Directed Against FACTOR VIII, Administered Intravenously in Healthy Male Volunteers.
Brief Title: A Phase I Study of Monoclonal Antibody TB-402 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Collaborators: BioInvent International AB (Industry)
Responsible Party: Geraldine Cahillane, ThromboGenics Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TB-402-001
Record Dates: First submitted 2008-01-09; First posted 2008-02-11 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Safety and tolerability
MeSH Terms: interventions — TB 402

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1 (Experimental)
  Interventions: Drug: TB-402
- 2 (Experimental)
  Interventions: Drug: TB-402
- 3 (Experimental)
  Interventions: Drug: TB-402
- 4 (Experimental)
  Interventions: Drug: TB-402
- 5 (Experimental)
  Interventions: Drug: TB-402
- 6 (Experimental)
  Interventions: Drug: TB-402
- 7 (Experimental)
  Interventions: Drug: TB-402
- 8 (Experimental)
  Interventions: Drug: TB-402
- 9 (Experimental)
  Interventions: Drug: TB-402
- 10 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TB-402 — Solution for infusion, 0.015ug/kg-1.8mg/kg, single dose, iv infusion over 30 minutes
  Arms: 1; 2; 3; 4; 5; 6; 7; 8; 9
Drug: Placebo
  Arms: 10

SUMMARY:
Dose escalation study to assess the safety and tolerability of TB-402, a monoclonal antibody directed against FVIII, versus placebo in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 45 (Groups 1-9) or 55 to 75 (Group 10) years of age
* No clinically important abnormal physical, laboratory, ECG findings
* Normal (or abnormal but ncs) supine blood pressure (BP) and heart rate (HR)

Exclusion Criteria:

* Self or family history of cardiovascular or pulmonary disorder, coagulation or bleeding disorders or reasonable suspicion of vascular malformations eg cerebral haemorrhage, aneurysm or premature stroke.
* Any autoimmune disease.
* Previous allergic reaction to immunoglobulin.
* Present, or history of, severe allergy, for example asthma or anaphylactic reactions or allergy requiring treatment.
* Consumption of aspirin, other non-steroidal anti-inflammatory drugs or other drugs known to affect platelet function or any other aspect of coagulation within 14 days before drug administration.
* Abnormal platelet function or clinically significant out of range values for any coagulation tests.
* History of important bleeding episodes eg haematemesis, rectal bleeding, severe or recurrent epistaxis, haemoptysis, haematuria or intracranial haemorrhage.
* Screening FVIII:C < 50%.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Jensen, M.D., Principal Investigator — Cyncron Clinical Research Unit
Locations (1):
- Cyncron Clinical Research Unit, Copenhagen, Denmark

REFERENCES:
- [Derived] Verhamme P, Pakola S, Jensen TJ, Berggren K, Sonesson E, Saint-Remy JM, Balchen T, Belmans A, Cahillane G, Stassen JM, Peerlinck K, Glazer S, Jacquemin M. Tolerability and pharmacokinetics of TB-402 in healthy male volunteers. Clin Ther. 2010 Jun;32(6):1205-20. doi: 10.1016/j.clinthera.2010.06.012. PMID 20637972